CLINICAL TRIAL: NCT07195877
Title: Real-life Assessment of the Safety and Performance of the "Infinite-Thread®" Permanent Tensor Thread on the Face, From the Thread & Lift Laboratory
Brief Title: Real-life Assessement of Safety and Perofmance of the of the "Infinite-Thread®" Permanent Tensor Thread
Status: Recruiting | Type: Observational
Sponsor: Thread and Lift (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: FILS-TENSEURS; 2024-A02819-38 (Other: ANSM)
Record Dates: First submitted 2025-08-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Face Tissue Elevation
Keywords: Tissue elevation; Infinite-Thread; Face; Aesthetic; Infinite-Thread®; permanent tensor thread; Thread&Lift
MeSH Terms: conditions — Facies | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Insertion/placement of tension threads — * Standard preoperative anti-staphylococcal antibiotic prophylaxis by intramuscular injection.
  * Disinfection of the surgical area.
  * Marking of the paths of the threads to be implanted according to the physician's choice.
  * Placement of sterile surgical drapes.
  * Local anesthesia of the paths.
  * Implantation of a needle (manufactured by Thread & Lift) and pulling of the threads into the subcutaneous tissue. Adjustment of the tension of all the implanted threads. Cutting of the ends of the threads.

SUMMARY:
The purpose of this post-market clinical follow-up is to assess the safety and performance of the "Infinite-Thread®" Permanent Tensor Thread on the Face. The study will assess the safety result up to 5 years after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 years or older
* Subject informed and not opposed to participating in the study
* Subject to be implanted with at least one Infinite-Thread® tension thread
* Person affiliated with a heallth care system/inssurance

Exclusion Criteria:

* Pregnant or breastfeeding women
* Contraindications (allergy to components, infection, systemic diseases)
* Subject prones to chronic pain
* Person deprived of liberty, under guardianship/curatorship, or under judicial protection
* Subject refusing to commit to not resorting to the following procedures during the 5 years following their intervention: Surgical facelift, Deep phenol peel, CO2 laser resurfacing & Lipofilling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject aged 18 years old or more who need of facial tissue enhancement.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess medical device safety at 5 years after intervention. | at 5 years follow-up
  The rate of sequelae and complications related to the device or procedure within 5 years after the intervention

SECONDARY OUTCOMES:
To assess the effectiveness of the Infinite-Thread® permanent tension thread by the subject (overall and by area) | At 3-months, 1,2,3,4 and 5 years follow-up
  Completion of effectiveness score by patient (GAIS) (overall and by area). It's a 5 points scale (1 to 5). The minimum value is 1 associated to a significant improvement and the maximum value is 5 associated to significant deterioration/worse.
To assess the effectiveness of the Infinite-Thread® permanent tension thread by the physician (overall and by area) | At 3-months, 1,2,3,4 and 5 years follow-up
  Completion of effectiveness score by physician (GAIS) (overall and by area). It's a 5 points scale (1 to 5). The minimum value is 1 associated to a significant improvement and the maximum value is 5 associated to significant deterioration/worse.
To assess the effectiveness of the Infinite-Thread® permanent tension thread by area by the physician. | At 3 months, 1, 2, 3, 4, and 5 years follow-up
  Physician effectiveness scale (5-point ordinal scales) by area. Values range from 0 to 4. 0 is the minimum value and the best (Non-sagging or non-marked area). 4 is the maximum and the worse value (Area that is significantly sagging or marked).
To assess the effectiveness of the Infinite-Thread® permanent tension thread by the independant assessor (physician) (overall and by area). | At 3-months, 1,2,3,4 and 5 years follow-up
  Completion of effectiveness score by independant assessor (physician) (GAIS) (overall and by area). Blind analysis of picture.
  It's a 5 points scale (1 to 5). The minimum value is 1 associated to a significant improvement and the maximum value is 5 associated to significant deterioration/worse.
To assess the effectiveness of the Infinite-Thread® permanent tension thread by area by the independent assessor (physician). | At 3 months, 1, 2, 3, 4, and 5 years follow-up
  Independent assessor (physican) effectiveness scale (5-point ordinal scales) by area. Blind analysis of picture.
  Values range from 0 to 4. 0 is the minimum value and the best (Non-sagging or non-marked area). 4 is the maximum and the worse value (Area that is significantly sagging or marked).

CONTACTS AND LOCATIONS:
Locations (1):
- Evamed/1Med, Hérouville-Saint-Clair, France

IPD SHARING:
Plan to Share IPD: No